CLINICAL TRIAL: NCT05144568
Title: The Effect of Nutrition Education on Premenstrual Syndrome: Randomized Controlled Study
Brief Title: The Effect of Nutrition Education on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Duygu MATARACI DEĞİRMENCİ, research assistant, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: orduüniversitesiDuyguMataracı1
Record Dates: First submitted 2021-10-18; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome; nutritional status; nutrition education; nursing students; university students
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Nutrition education will be given to participants with PMS in the experimental group.
  Interventions: Other: Nutrition education
- Control group (No Intervention)

INTERVENTIONS:
Other: Nutrition education — Nutrition education will be given to improve PMS
  Arms: experimental group

SUMMARY:
The aim of our study is to examine the effect of nutritional education given to university students with premenstrual syndrome (PMS) on premenstrual symptom severity, nutrient intake and anthropometric measures. Our hypothesis is that nutrition education reduces symptoms in students with PMS. The effect of nutrition education on premenstrual syndrome was evaluated. The sample for this study included 83 female students, with 43 in the experimental and 40 in the control group, who were studying at the health sciences faculty of a state university and met the inclusion criteria. Experimental and control groups were formed by randomized method. Nutrition training was given to the experimental group. Participant data were collected before and four months after nutrition training. The data were collected with the personal information form, Premenstrual Syndrome Scale and food consumption record form. Nutrient amounts were determined in the Nutrition Information System (BEBİS) program.

DETAILED DESCRIPTION:
1. INTRODUCTION Premenstrual Syndrome (PMS) is a condition in which physical, psychological and emotional symptoms related to the menstrual cycle of women are seen together. These symptoms experienced by many women occur before menstruation and disappear with menstrual bleeding. Imbalance in estrogen and progesterone levels, stress and malnutrition are among the factors affecting PMS.

   PMS, which has many symptoms such as changes in appetite, increased body weight, abdominal pain, back pain, headache, breast swelling and sensitivity, irritability, and fatigue, has incidence in Turkey in the range of 58.1% to 91.8%. It is known that individuals who do not exercise regularly, eat too much salt and sugar, and have high stress levels experience more PMS symptoms. While the presence of PMS in women causes an increase in health expenditures, loss of labor and low quality of life, in addition to these, it causes low concentration, absenteeism from school and academic failure.

   The etiology of premenstrual syndrome is not fully known, but one of the most emphasized reasons is hormone imbalance. Since the pathophysiology of PMS is not known exactly, the aim is to alleviate the severity of the symptoms during treatment of this syndrome. Non-pharmacological treatment methods such as exercise and diet are used. Studies reported that there is a positive relationship between increasing body mass index (BMI) and the risk of PMS. The incidence and severity of PMS is accepted to increase with simple carbohydrate consumption, and the aim is to reduce simple carbohydrate consumption and increase complex carbohydrate and fiber consumption in the treatment of PMS. It is reported that the consumption of foods with high fat content is a diet that increases the severity of PMS. Excessive consumption of salt, sugar, caffeine and alcohol negatively affects PMS.

   Studies conducted so far revealed various causes of PMS, and the effect of malnutrition on the etiology of PMS was mentioned. However, there are a few studies on providing nutrition training to individuals with PMS. Studies were conducted to show that excessive consumption of certain foods such as salt, sugar and caffeine, and insufficient intake of calcium, magnesium, B group vitamins and many other nutrients increase the severity of PMS. However, studies to reduce the severity of PMS by providing nutrition training to women with PMS are limited. This study was carried out to examine the effect of nutritional education given to nursing students studying at university on premenstrual symptom severity, nutrient intake and anthropometric measures.

   Research hypotheses:

   H1: Nutrition education has an impact on anthropometric measurements. H2: Nutrition education affects nutrient intake. H3: Nutrition education is effective in reducing the severity of premenstrual syndrome
2. METHODS 2.1. Participants and Recruitment The population of this randomized controlled experimental study consisted of 117 female students who scored 111 and higher on the premenstrual syndrome scale (PMSS). The sample of the study included 83 nursing students, 43 in the experimental group and 40 in the control group, who agreed to participate in the study and were eligible for the inclusion criteria. The groups were created using the randomization technique, and a computer program was used for randomization (https://www.randomizer.org/). The rate of participation in the research was 71%. Female students who volunteered to participate in the study, who had regular menstrual cycles and were over 18 years old were included in the study. Students with chronic disease, dieting in the last 3 months and using oral contraceptives were excluded from the study.

The reason for conducting the study with female students is to minimize confounding factors such as pregnancy, lactation, and the use of oral contraceptives.

2.2. Study Design The first data in the study were collected between June 3 and June 10, 2019 with a questionnaire prepared by the researchers, the Premenstrual Syndrome Scale, and a 24-hour retrospective food consumption record. After the first evaluation, nutrition training was given to the experimental group, and no intervention was made to the control group. Anthropometric measurements of the participants and a 24-hour retrospective food consumption record were completed again 4 months after the nutrition training (between September 23 and September 30, 2019) and PMSS was re-applied. With the information obtained, the effect of nutrition education on anthropometric measurements, daily nutrients and premenstrual symptom severity was examined.

2.3. Instruments 2.3.1. Question form. In the questionnaire, there were questions about the students' age, class of education, current place of residence, anthropometric measurements including body weight, height, waist and hip circumference, smoking status, exercise status, coffee and salt consumption, skipping meals status, skipped meals, reason for skipping meals and what they consumed in the last 24 hours.

2.3.2. Anthropometric measurements. Anthropometric measurements including body weight, height, waist and hip circumference of the participants were taken. Participant weight was measured with a portable digital scale in light clothing and without shoes, and height without shoes was measured with the aid of a meter fixed to the wall with the feet side by side and on the head Frankfort plane. For the waist circumference measurement, the midpoint of the lowest rib of the individual and the crista iliac crest were found and the circumference passing through the midpoint was measured with an inelastic tape measure. Hip circumference was measured with a non-stretch tape measure at the highest point of the hip circumference, standing by the side of the participant. BMI was calculated by the ratio of body weight in kg to the square of height in meters.

2.3.3. Premenstrual syndrome scale. The Premenstrual Syndrome Scale (PMSS), developed by Gençdoğan20 based on DSM-III and DSM-IVR criteria, consists of 44 questions. The PMSS is Likert type and its items are scored between 1 and 5 points. Lowest points of 44 and highest points of 220 can be obtained on the PMSS. The scale has a total of 9 subscales: depressive feeling, anxiety, fatigue, irritability, depressive thoughts, pain, changes in appetite, changes in sleeping habits and swelling. A higher score on the scale indicates that the severity of premenstrual syndrome is high. When the score of the total PMSS and subscales is higher than 50% of the total score, it is considered to indicate PMS. In the original study, the Cronbach alpha value for the whole scale was 0.75, in this study the Cronbach alpha value was 0.90 before nutrition education and 0.96 after the education. For premenstrual syndrome subscales, the Cronbach alpha values before and after the intervention were depressive feeling 0.85-0.89, anxiety 0.77-0.86, fatigue 0.81-0.87, irritability 0.88-0.92, depressive thoughts 0.82-0.91, pain 0.74-0.79, changes in appetite 0.55-0.58, changes in sleeping habits 0.77-0.79 and swelling 0.85-0.81.

2.4. Intervention-Nutrition Education In the experimental group, 43 students were divided into 4 groups, and each group received an hour of nutrition education. The education was carried out in classrooms where the students were trained, supported by a power point presentation. Nutritional sources of nutrients were taught, the relationship of some specific foods such as salt and coffee with premenstrual syndrome, the number of meals, meal time and importance of body weight control in premenstrual syndrome were emphasized. On the 30th and 60th days after the nutrition education, an e-mail was sent to the participants to inform them about nutrition in order to reinforce the education.

2.5. Ethical Issues Before starting the study, permission was obtained from Gençdoğan to use the PMS scale. In order to conduct the research, permission of the institution was obtained from Ordu University where the research was conducted (decision dated 26 April 2019 and numbered ….). Ethics committee approval was obtained from Ordu University Non-Interventional Clinical Research Ethics Committee (May 23, 2019 and numbered 2019/82). After the participants were informed about the study, their informed written consent was obtained. In this study, the principles of the Declaration of Helsinki were followed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* be woman
* have a regular menstrual cycle
* be 18 years or older

Exclusion Criteria:

* have a chronic illness
* have been on a diet in the last 3 months
* using oral contraceptives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is a study only on women with menstrual cycles. It is a study aimed at reducing the symptoms seen before the menstrual cycle. Therefore, the study was conducted with female participants.
Enrollment: 83 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of the nutrition education given to the experimental group was evaluated with the Premenstrual Syndrome Scale. | 3 months
  The Premenstrual Syndrome Scale consists of 44 questions. The PMSS is Likert type and its items are scored between 1 and 5 points. Lowest points of 44 and highest points of 220 can be obtained on the PMSS. The scale has a total of 9 subscales: depressive feeling, anxiety, fatigue, irritability, depressive thoughts, pain, changes in appetite, changes in sleeping habits and swelling. A higher score on the scale indicates that the severity of premenstrual syndrome is high. When the score of the total PMSS and subscales is higher than 50% of the total score, it is considered to indicate PMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No